CLINICAL TRIAL: NCT06494280
Title: Impact of Programmed Intermittent Epidural Bolus Compared With Continuous Epidural Infusion on Breakthrough Pain Among Laboring Nulliparous Women. A Randomized Controlled Trial
Brief Title: PIEB Compared With CEI on Breakthrough Pain in Nulliparous Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Holy Family Hospital, Nazareth, Israel (Other)
Responsible Party: Principal Investigator, Raed Salim, MD, head of obstetrics and gynecology department, Holy Family Hospital, Nazareth, Israel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 297\2024 HFH
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Breakthrough Pain
Keywords: Nullipara; Term pregnancy; Singleton; Vertex presentation; Latent phase; Maternal request for epidural; Visual analogue scale > 4
MeSH Terms: conditions — Breakthrough Pain | interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Active Comparator): Epidural analgesia will be maintained by receiving programmed intermittent 10ml bolus of 0.1% Bupivacaine and 2microgram\ml Fentanyl every one hour, until the delivery is completed, and lacerations are sutured.
  Interventions: Drug: programmed intermittent Bolus epidural analgesia
- control group (Active Comparator): Epidural analgesia will be maintained by receiving 10ml\h continuous infusion of 0.1% Bupivacaine and 2microgram\ml Fentanyl until the delivery is completed, and lacerations are sutured.
  Interventions: Drug: continuous epidural infusion

INTERVENTIONS:
Drug: programmed intermittent Bolus epidural analgesia — About 30 minutes after the end of the epidural and administration of the loading dose, the woman will be asked to report her pain level. If the VAS score <30, the woman will receive the study group protocol for pain maintenance, i.e., a programmed intermittent bolus of 10 ml of 0.1% bupivacaine and 2 μg/ml fentanyl every hour until the completion of labor and suturing of the incision. The participant can add to herself 5 ml of the same solution of Bupivacaine and Fentanyl every 30 minutes. The maximum dose that the parturient is allowed to receive is 20 ml for one hour.
  If a breakthrough pain appears during labor, a bolus of 10 ml of anesthetic solution with the same concentration will be added.
  Participants with a VAS score >30 after 30 minutes of the loading dose will be asked to perform a new epidural (if it was decided that the epidural failed) otherwise her data will not be collected for the final analysis of the study.
  Other Names: Bupivacaine + Fentanyl
  Arms: study group
Drug: continuous epidural infusion — About 30 minutes after the end of the epidural and administration of the loading dose, the woman will be asked to report her pain level. If the VAS score <30, the woman will receive the control group protocol for pain maintenance, i.e., 0.1% Bupivacaine and 2 μg/ml fentanyl as a continuous infusion per one hour, until the delivery is completed, and laceration is sutured. The participant can add to herself 5 ml of the same solution of Bupivacaine and Fentanyl every 30 minutes. The maximum dose that the parturient is allowed to receive is 20 ml for one hour.
  If a breakthrough pain appears during labor, a bolus of 10 ml of anesthetic solution with the same concentration will be added.
  Participants with a VAS score >30 after 30 minutes of the loading dose will be asked to perform a new epidural (if it was decided that the epidural failed) otherwise her data will not be collected for the final analysis of the study.
  Other Names: Bupivacaine + Fentanyl
  Arms: control group

SUMMARY:
The goal of this randomized controlled trial is to examine the impact of programmed intermittent bolus epidural analgesia technique on the incidence of breakthrough pain during labor in nulliparous women compared to continuous epidural infusion.

Nulliparous women will randomly be divided during labor into two groups; study group will receive mix of Bupivacaine and fentanyl once (bolus) every 60 minutes; the control group will receive continuously the same dose during an hour, until delivery.

DETAILED DESCRIPTION:
There are several pharmacological and non-pharmacological techniques for pain relief during labor. Epidural analgesia is considered the most effective modality for intrapartum pain relief.

Maintenance of epidural analgesia is achieved by different techniques; continuous epidural infusion (CEI), intermittent epidural analgesia (IEA), patient control epidural analgesia (PCEA) and combination between the techniques.

Another technique, the Programmed Intermittent Bolus Epidural Analgesia (PIBEA). The advantage of this technique is that boluses are given all the time at planned intervals, so laboring women do not depend on the medical staff to receive the bolus when there is a breakthrough pain.

This method has been reported to be associated with less motor block, lower incidence of instrumental vaginal deliveries, and less consumption of anesthetic agents when compared to CEI. There are no conclusive data regarding the use of PIBEA in combination with PCEA compared to CEI and PCEA on the effect of pain relief during labor and birth outcomes. The hypothesis of the current trial is that PIBEA and PCEA will decrease the incidence of breakthrough pain, and probably shorten the second stage of labor, lead to fewer instrumental deliveries and higher women's satisfaction compared to CEI and PCEA.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* Term pregnancy
* Singleton
* Vertex presentation
* Latent phase (cervical dilatation <6 cm)
* Epidural analgesia request
* Visual Analogue Scale score > 40

Exclusion Criteria:

* Estimated fetal weight > 4 kg
* Intra uterine fetal death
* Drug sensitivity
* Anomalous fetus
* Contraindication for epidural analgesia

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
breakthrough pain | 48 hours
  Incidence of breakthrough pain, defined as Visual Analogue Scale (VAS) score > 30.
  The VAS consists of a 100cm line, with two end points representing 0 ('no pain') and 100 (severe pain).

SECONDARY OUTCOMES:
manual bolus (top up) | 48 hours
  Number of participants who will require top up of Bupivacaine and Fentanyl due to breakthrough pain.
Hourly visual analogue scale | 48 hours
  Hourly pain according to visual analogue scale (VAS) score. The VAS consists of a 100cm line, with two end points representing score 0 (no pain) and score 100 (severe pain).
Time to delivery | 48 hours
  Time from epidural analgesia to delivery.
Oxytocin augmentation | 48 hours
  Incidence of women who will require Oxytocin for labor augmentation
Duration of second stage | 48 hours
  The time from complete cervical dilatation until delivery of the fetus (minutes)
Intrapartum fever | 48 hours
  Number of patients that will have intrapartum fever ≥ 38 °C
Number of patients that will require use of intrapartum use of antibiotic treatment. | 48 hours
  Number of patients that will require use of intrapartum use of antibiotic treatment due to intrapartum infection.
Mode of delivery | 48 hours
  Whether the birth was a normal spontaneous birth, operative vaginal birth or a cesarean section.
Indications for cesarean or operative vaginal deliveries | 48 hours
  Was the reason for operative vaginal delivery or cesarean delivery due to non-progressive labor, fetal status, or a combination of both?
duration of third stage | 48 hours
  time from delivery of the fetus the delivery of the placenta (minutes)
Early postpartum hemorrhage (PPH) | 48 hours
  Number of Participants with develop PPH
Hemoglobin level | 96 hours
  The lowest postpartum Hemoglobin level
Blood transfusion | 72 hours
  Number of Participants that will need blood transfusion.
Obstetric anal sphincter injury | 48 hours
  Number of Participants with that will develop 3rd and 4th degrees perineal lacerations.
Motor block of any leg | 48 hours
  Incidence of motor block will be assessed according to Bromage score:
  Bromage 0 = No motor block. Bromage 1 = the participant is unable to flex her hip Bromage 2 = the participant is able to flex her ankle but unable to flex her hip and knee Bromage 3 = the participant is unable to flex her hip, knee and ankle
Urinary retention | 48 hours
  Participant will not be able to urinate spontaneously 6 hours after delivery
Dural puncture | 48 hours
  Incidence of dural puncture during performing epidural analgesia
Side effects related epidural analgesia use | 48 hours
  nausea, vomiting, and pruritis
mean arterial blood pressure | 48 hours
  mean arterial blood pressure (mmHg) of the participant during labor
systolic blood pressure < 90mmHg | 48 hours
  incidence of systolic blood pressure < 90 during labor
Bupivacaine consumption | 48 hours
  total Bupivacaine consumption during labor (ml)
maternal satisfaction | 48 hours
  participant satisfaction from labor experience from 1 to 10.
  1= very dissatisfied 10 = very satisfied
Apgar score (0 to 10) | 48 hours
  APGAR< 7 after 1 and 5 minutes where lower scores mean a worse outcome.
fetal cord artery pH | 48 hours
  Cord artery pH <7.1
meconium staining | 48 hours
  Incidence of meconium-stained amniotic fluid before delivery of the fetus
Neonatal sepsis | 72 hours
  Incidence of early neonatal sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Raed Salim, MD, Study Chair — Holy Family Hospital, Nazareth, Israel
Locations (1):
- Holy Family Hospital, Nazareth, Israel

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after publication
Access Criteria: Access to IPD can be requested by qualified researchers and will be granted after review and approval of a research proposal and statistical analysis plan and execution of a data sharing agreement.
  For more information or to apply, please contact the Principal Investigator

REFERENCES:
- [Result] 1. American College of Obstetricians and Gynecologists. Obstetric analgesia and anesthesia. ACOG Practice Bulletin No. 209. Obstet Gynecol. 2019;133:e208-25. 2. Anim-Somuah M, Smyth RM, Cyna AM, Cuthbert A. Epidural versus non-epidural or no analgesia for pain management in labour. Cochrane Database of Systematic Reviews 2018:5;CD000331. 3. Jones L, Othman M, Dowswell T, Alfirevic Z, Gates S, Newburn M, et al. Pain management for women in labour: an overview of systematic reviews. Cochrane Database of Systematic Reviews 2012:3;CD009234. 4. George RB, Allen TK, Habib AS. Intermittent epidural bolus compared with continuous epidural infusions for labor analgesia: a systematic review and meta-analysis. Anesth Analg 2013;116:133-44. 5. Sng BL, Zeng Y, de Souza NNA, Leong WL, Oh TT, Siddiqui FJ, Assam PN, Han NR, Chan ES, Sia AT. Automated mandatory bolus versus basal infusion for maintenance of epidural analgesia in labour. Cochrane Database Syst Rev. 2018;5:CD011344. 6. Ferrer LE, Romero DJ, Vasquez OI, Matute EC, Van de Velde M. Effect of programmed intermittent epidural boluses and continuous epidural infusion on labor analgesia and obstetric outcomes: a randomized controlled trial. Arch Gynecol Obstet. 2017;296:915-22. 7. Ojo OA, Mehdiratta JE, Gamez BH, Hunting J, Habib AS. Comparison of programmed intermittent epidural boluses with continuous epidural infusion for the maintenance of labor analgesia: a randomized, controlled, double-blind study. Anesth Analg. 2020;130:426-35. 8. Haidl F, Arne Rosseland L, Rorvik AM, Dahl V. Programmed intermittent boluses vs continuous epidural infusion in labor using an adrenaline containing solution: A randomized trial. Acta Anaesthesiol Scand. 2020;64:1505-12. 9. Riazanova OV, Alexandrovich YS, Guseva YV, Ioscovich AM. A randomized comparison of low dose ropivacaine programmed intermittent epidural bolus with continuous epidural infusion for labour analgesia. Rom J Anaesth Intensive Care. 2019;26:25-30. 10. Fan Y, Hou W, Feng S, Mao P, Wang X, Jiang J, Yuan H, Shen X, Feng S, Li P. Programmed intermittent epidural bolus decreases the incidence of intra-partum fever for labor analgesia in primiparous women: a randomized controlled study. Arch Gynecol Obstet. 2019;300:1551-7 11. Xu J, Zhou J, Xiao H, Pan S, Liu J, Shang Y, Yao S. A systematic review and meta-analysis comparing programmed intermittent bolus and continuous infusion as the background infusion for parturient-controlled epidural analgesia. Sci Rep. 2019;9:2583. 12. Wang XX, Zhang XL, Zhang ZX, Xin ZQ, Guo HJ, Liu HY, Xiao J, Zhang YL, Yuan SZ. Programmed intermittent epidural bolus in parturients: a meta-analysis of randomized controlled trials. Medicine (Baltimore). 2022;101: e28742. 13. Bullingham A, Liang S, Edmonds E, Mathur S, Sharma S. Continuous epidural infusion vs programmed intermittent epidural bolus for labour analgesia: a prospective, controlled, before-and-after cohort study of labour outcomes. Br J Anaesth. 2018;121:432-7. 14. Lin Y, Li Q, Liu J, Yang R, Liu J. Comparison of continuous epidural infusion and programmed intermittent epidural bolus in labor analgesia. Ther Clin Risk Manag. 2016;12:1107-12. 15. Lim Y, Sia AT, Ocampo C. Automated regular boluses for epidural analgesia: a comparison with continuous infusion. Int J Obstet Anesth. 2005;14:305-9. 16. Salim R, Nachum Z, Moscovici R, Lavee M, Shalev E. Continuous compared with intermittent epidural infusion on progress of labor and patient satisfaction. Obstet Gynecol 2005;106:301-6. 17. Lim Y, Ocampo CE, Supandji M, Teoh WH, Sia AT. A randomized controlled trial of three patient-controlled epidural analgesia regimens for labor. Anesth Analg 2008;107:1968-72. 18. Capogna G, Camorcia M, Stirparo S, Farcomeni A. Programmed intermittent epidural bolus versus continuous epidural infusion for labor analgesia: the effects on maternal motor function and labor outcome. A randomized double-blind study in nulliparous women. Anesth Analg 2011;113:826-31. 19. Carvalho B, George RB, Cobb B, McKenzie C, Riley ET. Implementation of Programmed Intermittent Epidural Bolus for the Maintenance of Labor Analgesia. Anesth Analg 2016;123:965-71 20. Diez-Picazo LD, Guasch E, Brogly N, Gilsanz F. Is breakthrough pain better managed by adding programmed intermittent epidural bolus to a background infusion during labor epidural analgesia? A randomized controlled trial. Minerva Anestesiol. 2019;85:1097-104. 21. Roofthooft E, Barbé A, Schildermans J, Cromheecke S, Devroe S, Fieuws S, Rex S, Wong CA, Van de Velde M. Programmed intermittent epidural bolus vs. patient-controlled epidural analgesia for maintenance of labour analgesia: a two-centre, double-blind, randomised study. Anaesthesia. 2020;75:1635-42. 22. Sultan P, Murphy C, Halpern S, Carvalho B. The effect of low concentrations versus high concentrations of local anesthetics for labour analgesia on obstetric and anesthetic outcomes: a meta-analysis. Can J Anaesth. 2013;60:840-54.